CLINICAL TRIAL: NCT06452303
Title: The Patient Cohort for Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hua Meng, Director of the General Surgery Department & Obesity and Metabolic Disease Center of China-Japan Friendship Hospital, China-Japan Friendship Hospital
Other Study IDs: PCBS
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Height, Weight, Waist Circumference, Hip Circumference; Preoperative Laboratory Examination Status; Preoperative Routine Examination Results; Laboratory and Examination Results During Follow-up
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is based at the National Integrated Traditional Chinese and Western Medicine Medical Center and leverages the centralized strengths of our department, which integrates multiple disciplines (general surgery, endocrinology, nutrition, exercise, and traditional Chinese medicine). It focuses on key scientific issues in the comprehensive management of bariatric surgery throughout the entire treatment cycle. By recording key indicators of patients before and after surgery and using methods such as machine learning to predict postoperative complications, we aim to enhance precision management. Ultimately, we will establish a refined diagnosis and treatment system for metabolic weight loss surgery, promote its application, and thereby raise the standardized management level of weight loss and metabolic disciplines in our hospital and primary care units nationwide. This will improve patient outcomes and reduce the healthcare burden.

ELIGIBILITY:
Inclusion Criteria:

* 1、For those with simple obesity, BMI ≥ 32.5, or 27.5 ≤ BMI < 32.5, who have difficulty controlling their condition with lifestyle modifications and medical treatment, and who meet at least two criteria for metabolic syndrome components, or have comorbidities.

  2、For those with simple obesity, 27.5 ≤ BMI < 32.5, and with male waist circumference ≥ 90 cm, female waist circumference ≥ 85 cm, and imaging studies suggesting central obesity.

  3、For those with type 2 diabetes, BMI ≥ 27.5, who still have some residual insulin secretion capacity.

Exclusion Criteria:

* 1、Non-obese type 1 diabetes; 2、Those for whom the purpose of treatment is T2DM, but whose pancreatic beta-cell function is largely lost, with a BMI < 25.0; 3、Age < 16 years or age > 65 years; 4、Pregnant women with diabetes and patients with certain special types of diabetes; 5、Those with a cognitive disorder or immature intelligence, and who cannot control their behavior; 6、Those whose expectations for the surgery are not realistic; 7、Those unwilling to assume the risks of potential surgical complications; 8、Those unable to comply with postoperative dietary and lifestyle changes, showing poor compliance; 9、Those in poor general health, who are unable to tolerate general anesthesia or surgery.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals planning to undergo bariatric surgery in China-Japan Friendship Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
weight | Before bariatric surgery, 1 month after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China